CLINICAL TRIAL: NCT06077825
Title: Does Symmetrical Lower Limb Loads Distribution Effects Balance and Risk of Fall After Total Hip Arthroplasty?
Brief Title: Effects of Lower Limbs Symmetrical Loading on Risk of Fall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Burcu Özdemir Kocabey, PhD, Bahçeşehir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AcibademHospital
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Total Hip Replacement
Keywords: total hip arthroplasty; static balance; postoperative rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): 30 patients who underwent total hip arthroplasty surgery took part in the experimental group.
  Interventions: Other: postoperative rehabilitation

INTERVENTIONS:
Other: postoperative rehabilitation — 30 patients took postoperative rehabilitation after total hip arthroplasty surgery, 3 times a week, for 6 weeks. They took conventional rehabilitation (hip range of motion exercises, progressive strengthening exercises for hip and knee muscles, balance and proprioceptive exercises and gait training).

SUMMARY:
Objective: To assess the impact of total hip arthroplasty (THA) on functional outcomes and fall risk in patients with hip osteoarthritis. The objective was to investigate the effectiveness of physical therapy in postoperative rehabilitation and identify fall risk factors to guide fall prevention strategies after THA.

Methods: A non-randomized, interventional clinical trial was conducted with 30 patients scheduled for THA. Functional outcomes were evaluated using the Harris Hip Score (HHS), 40-meter fast-paced walk test (40mFPWT), 30-Second Chair Test, and Western Ontario McMaster Universities Osteoarthritis Index (WOMAC). Balance and fall risk were assessed using the Single-Leg Standing Test and a posturography device (TETRAX). The Nottingham Health Profile (NHP) was used to measure subjective health status and quality of life. Assessments were performed preoperatively, at 6 weeks postoperatively, and at 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiographic evidence of unilateral hip osteoarthritis
* Volunteering to participate in the study

Exclusion Criteria:

* History of neurologic disorders affecting postural control (e.g., Parkinson disease)
* Have other problems that affect balance, such as vertigo
* Undergoing revision hip surgery
* Osteoarthritis in the other lower extremity joints

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | preoperative, postoperative 6 weeks and 3 months
  min-max (0-100) Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
40-meter fast-paced walk test | preoperative, postoperative 6 weeks and 3 months
30-Second Chair Test | preoperative, postoperative 6 weeks and 3 months
Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | preoperative, postoperative 6 weeks and 3 months
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain, Stiffness, Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Static balance and fall risk | preoperative, postoperative 6 weeks and 3 months
  It was assessed with Posturography device (TETRAX)
Single-Leg Standing Test | preoperative, postoperative 6 weeks and 3 months

SECONDARY OUTCOMES:
The Nottingham Health Profile (NHP) | preoperative, postoperative 6 weeks and 3 months
  The NHP is composed of 38 items divided into six domains:
  1. Sleep
  2. Mobility
  3. Energy
  4. Pain
  5. Emotional reactions
  6. Social isolation Items use a Yes/No answer format. Each item is weighted. NHP scores are calculated by averaging domain scores. Total scores range from 0 (no perceived distress) to 100 (maximum perceived distress).

CONTACTS AND LOCATIONS:
Overall Officials: Selvi Yüce, PhD(c), Principal Investigator — Acibadem Maslak Hospital